CLINICAL TRIAL: NCT07331116
Title: Correlations Between Biopsy Verified Myocardial Fibrosis and Echocardiography Parameters in Patients With Severe Aortic Stenosis
Brief Title: Echocardiography Findings in Patients With Myocardial Fibrosis and Severe Aortic Stenosis
Acronym: SAS-fibrosis
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Rikshospitalet University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/1068b
Record Dates: First submitted 2025-10-01; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis; Myocardial Fibrosis
Keywords: Myocardial fibrosis; Endomyocardial biopsy; Echocardiography; Aortic stenosis; Diastolic dysfunction
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic stenosis with biopsy-verified myocardial fibrosis: Periopererative echocardiography
  Interventions: Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Cardiac magnetic resonance imaging
- Aortic stenosis without biopsy-verified myocardial fibrosis: Periopererative echocardiography
  Interventions: Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Transthoracic echocardiography, performed close in time to the endomyocardial biopsy taken during aortic valve replacement procedure
Diagnostic Test: Cardiac magnetic resonance imaging — Cardiac magnetic resonance imaging was taken on selected patients without contraindications. The CMR protocol was changed midway during study inclusions (May 2017), in order to better be able to quantify myocardial fibrosis.

SUMMARY:
Patients with aortic stenosis waiting for aortic valve repair were investigated with echocardiography preoperatively, and a myocardial biospy was taken during the operation. We aim to perform a retrospective analysis of these data, to look for correlations between biopsy-verified myocardial fibrosis and echocardiography parameters.

The patients also had cardiac magnetic resonance imaging performed, for a non-invasive quantification of myocardial fibrosis.

DETAILED DESCRIPTION:
The primary purpose of the study is to retrospectively compare echocardiography measurements with a myocardial biopsy taken perioperatively in patients with aortic stenosis requiring aortic valve replacement.

Echocardiography and endomyocardial biopsy have been performed in close proximity in time. Due to a small sample size and a large number of echocardiography measurements being possible, only a limited number of prespecified comparisons are performed.

Cardiac magnetic resonance (CMR) was also performed in patients without contraindication, providing a non-invasive gold standard for diffuse fibrosis and replacement fibrosis. A secondary goal will be to investigate how echocardiography parameters performs compared to CMR in quantifying myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Planned for aortic valve replacement for symptomatic, severe aortic stenosis

Exclusion Criteria:

* Previous myocardial infarction / coronary disease that can cause fibrosis
* Do not wish to participate in study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is retrospective. Study participants has been selected among patients on waiting list for aortic valve replacement at Ullevaal Hospital, Oslo, Norway. Ages between 18 and 80 years, with no known other cardiac condition that can cause myocardial fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Echocardiography parameters of systolic and diastolic function | The time between echocardiography exam and endomyocardial biopsy was kept as short as possible, and not more than one month apart. If no cardiac event had happened in between, we could now regard echocardiography and biopsy being taken at the same time.
  Echocardiograhic parameters on structure and function of the heart, as described in guidelines for echocardiography assessment:
  Basal hypertrophy of interventricular septum, in mm. LV end diastolic mass (preferably from 3D volume of LV) LV end diastolic mass, indexed (preferably from 3D volume of LV) Left ventricular global longitudinal strain (%) Left ventricular ejection fraction, 3D Left ventricular septal strain rate, peak systolic, sample placed in basal septum Grading of diastolic dysfunction (ref EACVI/ASE guidelines) Left atrial strain, reservoir function, biplane Left atrial strain, conduit function , biplane Left atrial strain, (atrial) contraction phase, biplane Severity of aortic stenosis, evaluated by echocardiography (mild, moderate, severe)

SECONDARY OUTCOMES:
CMR parameters of systolic and diastolic function | CMR was taken preoperatively, and at 1-year postoperative check-up
  Left ventricular (LV) end diastolic volume, CMR LV end systolic volume, CMR LV stroke volume, CMR LV ejection fraction, CMR LV cardiac output, CMR LV cardiac index, CMR Global peak wall thickness, CMR CMR-dreived left ventricular mass, in end-diastole
  Left atrial volume in left atrial end systole, measured with CMR (left ventricular ED) Left atrial volume in left atrial end diastole, measured with CMR (left ventricular ES) Left atrial ejecton fraction, measured with CMR
  Global native T1 in myocardium, CMR Global post contrast T1 in myocardium, CMR Global ECV value in myocardium, CMR

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almaas VM, Haugaa KH, Strom EH, Scott H, Smith HJ, Dahl CP, Geiran OR, Endresen K, Aakhus S, Amlie JP, Edvardsen T. Noninvasive assessment of myocardial fibrosis in patients with obstructive hypertrophic cardiomyopathy. Heart. 2014 Apr;100(8):631-8. doi: 10.1136/heartjnl-2013-304923. Epub 2013 Dec 24. PMID 24368281